CLINICAL TRIAL: NCT04365491
Title: European Society for Trauma and Emergency Surgery (ESTES) Cohort Study Snapshot Audit 2020 - Acute Appendicitis
Acronym: SnapAppy
Status: Completed | Type: Observational
Sponsor: Gary Alan Bass, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Gary Alan Bass, MD PhD, ESTES Cohort Studies Committee Chairperson, European Society for Trauma and Emergency Surgery
Organization: European Society for Trauma and Emergency Surgery (Other)
Other Study IDs: ESTESSnapshot2020Appendix
Record Dates: First submitted 2020-04-22; First posted 2020-04-28 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Acute appendicitis is an extremely common surgical emergency. Traditionally, appendicitis has been managed surgically. Recently, however, variability in management of acute appendicitis has emerged, with some clinicians practising conservative, i.e. non-operative, management in selected patients. This high-quality pan-European, prospective audit will establish current practices and correlate them against outcomes.

Aim To explore differences in patient presentation, clinical course and outcomes for acute appendicitis across international clinical Centres to identify areas of practice variability in the presentation, management and complications of acute appendicitis.

Endpoints A three-stage data collection strategy will be used in this audit. There will be a 90 day prospective period for data collection during a six month window from September 2020 to end February 2021. Data collection will consist of collecting patient demographics, details of management (conservative vs surgical) and outcomes. Several outcomes measures will be used, including surgical mortality, morbidity (Clavien-Dindo Grade 2 and above) and length of hospital stay.

The data collection points are as follows:

1. 90 Day Prospective Audit Collecting anytime during 6-month window:

   * Demographics
   * Operative technique
   * Use of antibiotics
   * Conservative vs surgical management
   * Outcomes
2. All eligible patients will be followed up to 90 days from their admission

   * Readmissions will be flagged and identified
   * Complications within the 90 day period will be recorded
3. Patients who have a complete data set at 90 days post presentation will be followed up to the 1-year mark • Incomplete data sets will be excluded from the study

Methods: This 90 day prospective audit will be performed across Europe from September 2020 to end February 2021., and will be co-ordinated by a designated committee of European Society of Trauma and Emergency Surgery. This will be preceded by a one-week, three-Centre pilot. Sites will be asked to pre-register for the audit and will be required to obtain appropriate regional or national approvals in advance of the enrolment date.

During the study period, all eligible patients with acute appendicitis will be recorded contemporaneously and followed-up through to 90 days from their admission. The audit will be performed using a standardised pre-determined protocol, instrument and a secure online database. The report of this audit will be prepared in accordance with guidelines set by the STROBE (strengthening the reporting of observational studies in epidemiology) statement for observational studies.

Discussion: This multi-centre, snapshot audit will be delivered by emergency surgeons and trainees in an coordinated and homogenous manner. The data obtained about areas of variability in provision or practice, and how this may impact upon outcomes, will serve to improve overall patient care as well as being hypothesis generating and inform areas needing future prospective study.

ELIGIBILITY:
6.4 Inclusion Criteria

Adult patients (≥16 years of age) admitted for:

Acute Appendicitis

Procedures which should be included:

1. Appendectomy (open, laparoscopic or robotic)
2. Diagnostic laparoscopy
3. Partial right hemicolectomy (for appendiceal mass or carcinoid tumour) Exclusion Criteria

   * Mesenteric adenitis
   * Ovarian pathology

Methods for identifying patients

Multiple methods may be used according to local circumstances/staffing:

1. Daily review of emergency department (non-operative) and operating room lists
2. Daily review of team handover sheets / emergency admission lists / ward lists
3. Review of operating room logbooks
4. Use of electronic systems to flag any readmissions of patients identified and treated

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All hospitals/units performing general surgery are eligible to join this audit. No unit size or case throughput stipulations are made. Countries outside Europe can also participate in this audit.
  All participating centres will register with the ESTES cohort study office and will be responsible for their own local approvals process prior to the start of the data collection period. Inclusion of data sets will be subject to local approval from participating clinical Centres.
  Normal patient follow-up pathways can be utilised to obtain outcomes data. No additional visits or changes to normal follow-up should be made. However, local investigators should be proactive in identifying post-diagnosis. These may include reviewing the patient notes (paper and electronic) during admission and before discharge to note in-hospital complications, reviewing hospital systems to check for re-attendances or re-admissions, and reviewing post-operative radiology reports.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of acute appendicitis | 3 months
  Incidence of acute appendicitis

OTHER OUTCOMES:
Post-operative (or non-operative complications) | 90 days
  Complications related to disease and/or therapies within 90 post operative days
Length of post-operative stay in the hospital | 90 days
cost-analysis of treatment | 90 days
Re-admission within 90 postoperative days | 90 days
Number of participants with histopathological results, differences in age and clinical presentation | 90 days
Time to surgery | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Eanna J Ryan, MD MRCSI, Study Director — St Vincent's University Hospital, Ireland; Shahin Mohseni, MD, PhD, Study Chair — Orebro University Hospital, Sweden; Gary A Bass, MD, MS, Principal Investigator — Dept Traumatology, Surgical Critical Care, University of Pennsylvania, Philadelphia, PA, USA
Locations (1):
- Tallaght University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Pooled Data will be published. Subgroup analyses by disease, technique or outcome variables may be presented, but no hospital-level or surgeon-level data will be published whereby an individual patient, unit or surgeon can be identified. If local investigators would like their own unit's raw data for benchmarking purposes and local presentation/discussion, this can be made available after the end of the study; however, it will not be possible to de-anonymise patient data stored in Smart-Trial, in strict compliance with GDPR.
  The ESTES Cohort Studies Committee welcomes the use of the data for further research that benefits patients. Data sharing is subject to ESTES approval and appropriate safeguarding. Future sub-projects must comply with our policy of single corporate authorship e.g. "ESTES Cohort Studies Group". Authors' contributions will be highlighted in accordance with the recommendations for the conduct, reporting, editing, and publication of scholarly work in medical journals.

REFERENCES:
- [Derived] Bass GA, Kaplan LJ, Forssten MP, Walsh TN, Cao Y, Mohseni S; ESTES SnapAppy Group. Techniques for mesoappendix transection and appendix resection: insights from the ESTES SnapAppy study. Eur J Trauma Emerg Surg. 2023 Feb;49(1):17-32. doi: 10.1007/s00068-022-02191-8. Epub 2023 Jan 24. PMID 36693948
- [Derived] Young N, Ahl Hulme R, Forssten MP, Kaplan LJ, Walsh TN, Cao Y, Mohseni S, Bass GA; ESTES SnapAppy Group. Graded operative autonomy in emergency appendectomy mirrors case-complexity: surgical training insights from the SnapAppy prospective observational study. Eur J Trauma Emerg Surg. 2023 Feb;49(1):33-44. doi: 10.1007/s00068-022-02142-3. Epub 2023 Jan 16. PMID 36646862